CLINICAL TRIAL: NCT04849663
Title: Comparative Evaluation of Buccal Fat Pad and Subepithelial Connective Tissue Graft in the Treatment of Localized Recession (Randomized Clinical Trial)
Brief Title: Comparative Evaluation of Buccal Fat Pad and Subepithelial Connective Tissue Graft
Acronym: RCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, shehad wael, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASU689
Record Dates: First submitted 2021-03-31; First posted 2021-04-19 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Use of free fat graft to cover exposed root
  Interventions: Biological: free fat graft
- control group (Active Comparator): use of sub epithelial connective tissue graft to cover exposed root
  Interventions: Biological: subepithelial graft

INTERVENTIONS:
Biological: free fat graft — fat harvested from patient will be used to cover exposed root
  Arms: study group
Biological: subepithelial graft — subepitheial graft harvested from palate
  Arms: control group

SUMMARY:
Compare between Buccal fat pad and subepithelial connective tissue graft in treatment of localized recession.

Primary objective: to evaluate root coverage in terms of gingival thickness and esthetic.

Secondary objective: to evaluate patient satisfaction and postoperative pain.

DETAILED DESCRIPTION:
Material and Methods

16 patients from outpatient Oral Diagnosis dental clinic will participate in this study.

Patient selection and hospitalization

Prospective randomized clinical trial will be conducted on patients requiring correction of gingival recession. The research will be reviewed by the ethical committee of Faculty of Dentistry Ain Shams University.

Patient Grouping

Patient will be randomly allocated into one of the two groups:

control group (8 patients): will be treated with coronally advanced flap combined with subepithelial Connective tissue graft (SCTG).

Study group(8 patients): will be treated with coronally advanced flap combined with buccal fat pad (BFP).

Preoperative Assessment

For all patients routine radiographic investigations are required. The first phase of therapy formed of oral hygiene measures, scaling, subgingival debridement and correction of any disturbance in occlusion needed. A periodontal evaluation should be done two weeks after phase I therapy.

A stent will be made for each defect with vertical groove located at the mid-labial region to standardize the placement and angulation of probe while taking measurement. All measurements will be taken with a standardized Williams graduated periodontal probe (Hu-Friedy).

Surgical procedure:

* Oral antiseptic mouthwash will be used before anaesthetizing the surgical area. A field block anesthesia at the surgical area is given with a lidocaine and epinephrine-containing solution.

  a) Recipient site preparation
* A split-thickness flap will be reflected by a horizontal incision made at the papilla base, mesial and distal to the recession defects. Two slightly divergent incisions will be released from the end of the previous horizontal incisions with a full-thickness flap starting from margin of the gingiva reaching 3-4 mm after the exposed bone then continue with a split-thickness extending to the alveolar mucosa .
* After flap elevation scaling, planing of the exposed root followed by root conditioning with a tetracycline solution (125 mg tetracycline/ml of saline). In the study group sites, previously prepared BFP or a subepihelial CT graft in control group will be applied over the exposed root a single sling suture will fix the flap just coronal to the Cemento-enamel junction (CEJ). Flaps will also be coronally positioned.

  b) Donor site:
* In study group the buccal vestibule is anesthetized in vicinity of the first and second maxillary molar. The cheek will be retracted laterally and a mucosal incision will be made while leaving a cuff of non- attached mucosa for closure. The incision will be done throughout the mucosa and muscle meanwhile an external pressure will be applied on the skin in the area of the buccal fat pad. After the buccal fat pad exposure, the fascia is pierced with scissors. With a continuous external pressure on the cheeck a long hemostat is used to spread and manipulate the fat. With minimal delicate traction, the protruding portion of the fat pad is gently grasped and pulled outside of the incision then the fat is clamped at the base and the required amount is harvested and excised to be used in donor site. The incision is closed with suture .
* The control group will receive SCTG from the palate with a single incision technique .

Postoperatively patients will be covered by Augmentine 1 gm tablets every 12 hours and flagyl 500 mg every eight hours. Analgesics are given in a combined protocol; where ibuprofen 600mg and paracetamol 1gm are alternating. The patient is instructed to use 0.12% chlorhexidine mouthwash three times daily for two weeks.

Methods of assessment

The parameters which should be measured at baseline, 3 and 6 months after surgery:

1. Plaque index (PI) will be recorded according to Silness and Loe .
2. Gingival index (GI) will be recorded according to Loe and Silness .
3. Probing depth (PD).
4. Clinical attachment level (CAL).
5. Recession depth (RD).
6. Recession width (RW).
7. Percentage of mean root coverage (MRC %) will be calculated as ([RD preoperative - RD postoperative]/RD preoperative) × 100%.
8. Width of keratinized tissue (WKT).
9. Gingival thickness (GTH).
10. Root coverage esthetic score (RES).
11. Pain level will be assessed by verbal, numeric scale and by recording amount of analgesic intake postoperatively.

Result presentation and statistics

Results will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be above 18 years.
* Patient included in the study will be with Miller class II recession defect.
* Patient having at least 1 mm of residual keratinized tissue.

Exclusion Criteria:

* Patient with Systemic Problem affecting the results of periodontal Therapy.
* Patients having allergy to drugs.
* Pregnant women.
* Patients with any smoking habits.
* Patients having bleeding problems or on anticoagulant therapy.
* Patients having caries or restorations in relation to the treated site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
evaluation of root coverage esthetic score | 6 months
  evaluation of root gingival coverage after modified Coronally advanced flap the scale is from 1-4 ... based on degree of coverage the score will be given 1=1005, 2=75%, 3=50%, 4=25%

CONTACTS AND LOCATIONS:
Overall Officials: shehad wael, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No